CLINICAL TRIAL: NCT03495570
Title: An Observational Study Exploring the Utility of the Sysmex-XN 20 Analyser to Assess Lymphocyte Subsets and Other Haematological Parameters in Chronic or Acute Viral Infections,
Brief Title: Sysmex-XN 20 Analyser to Assess Lymphocyte Subsets and Other Haematological Parameters in Chronic/Acute Viral Infections
Acronym: SASA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: Central and North West London NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UCL 17/0634
Record Dates: First submitted 2018-03-21; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Diagnostic; Chronic Viral Hepatitis B; Chronic Hepatitis C; Chronic HIV Infection
Keywords: immunological
MeSH Terms: conditions — Disease; Hepatitis B, Chronic; Hepatitis C, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A: HIV-infected (chronic or acute infection) with a HIV viral load of >1000 copies/mL in the 6 months prior to study entry and not (yet) in receipt of combination antiretroviral therapy (cART) at study entry.
  Interventions: Diagnostic Test: blood draw
- B: HIV-infected on cART with HIV viral load <50 copies/mL within the 6 months prior to study entry, at least one measure of HCV (chronic or acute infection) showing a detectable HCV viral load and not in receipt of HCV treatment at study entry.
  Interventions: Diagnostic Test: blood draw
- C: HCV mono-infected (chronic or acute infection) with detectable HCV viral load (>lower limit of quantification) in the prior 6 months and not in receipt of HCV treatment at study entry.
  Interventions: Diagnostic Test: blood draw
- D: HBV mono-infected (chronic or acute infection) patients with detectable HBV viral load in the prior 6 months and not in receipt of HBV treatment at study entry.
  Interventions: Diagnostic Test: blood draw

INTERVENTIONS:
Diagnostic Test: blood draw — single one time blood draw to measure lymphocyte panels included activated lymphocytes using remnant sample from a full blood count
  Other Names: lymphocytes panels as measured by Sysmex XN-20 analyser

SUMMARY:
The XN-20, is a full blood count (FBC) analyser with an extended differential counting and flagging System. The XN-Series' individual channels allow real-time reflex analysis, and uses a two stage process to classify the white blood count (WBC) sub-populations and detect the presence of abnormal reactive and malignant cells. In regards to lymphocytes in the peripheral blood, the machine has the capacity to distinguish activated from non-activated T-cell subsets using a very small volume of EDTA sample (88uL) (including remnant sample from a standard full blood count) with results available in 1.5 minutes. It is a fully automated process and can be considered as an alternative rapid flow cytometry method.

Objective of the SASA study: to investigate the signal pattern of white blood cells assessed using the XN-20 full blood count platform in patients with untreated viral infections i.e. HIV, HCV and HBV. The data from the analysis will be reviewed in conjunction with patient's demographic and clinical disease characteristics with the aim of detecting characteristic cell populations that can be used in the development of system flags for future studies.

DETAILED DESCRIPTION:
Study design: observational pilot study. Approximately one hundred, participants (25 in each of group, A to D), will be enrolled at a single clinical site.

Study question: Do participants who have chronic or acute viral infections i.e. untreated HIV, HIV-HCV with treated HIV and untreated HCV, untreated HCV monoinfection or untreated HBV monoinfection, have a significant excess of activated lymphocytes as measured by D1+D2 on the XN WDF channel using the XN-20 analyser?

Objectives:

Primary: To assess whether participants who have chronic or acute viral infections have a significant excess of activated lymphocytes measured by the Sysmex-XN 20 analyser.

Secondary: To compare, the absolute numbers and percentages of lymphocytes subsets as measured in the Sysmex-XN 20 analyser to the percentages of these cells when measured using standard laboratory methods i.e. flow cytometry.

Primary Outcome Measure(s): Percentage of lymphocytes measured in area D1+D2 of the XN WDF and W1/W2 ratio from the WPC channel.

Secondary Outcome Measure(s ):

1. % lymphocytes in the D1 area of the XN WDF channel;
2. % lymphocytes in the D2 area of the XN WDF channel;
3. % lymphocytes in the D0 area of the XN WDF channel;
4. correlation between CD4+ T-cells (as measured by standard flow cytometry) and the D1+D2 area on the XN WDF channel;
5. correlation between CD8+ T-cells (as measured by standard flow cytometry) and the D1+D2 area on the XN WDF channel;
6. correlation between CD4+ T-cells (as measured by standard flow cytometry) and the W1/W2 area on the XN WPC channel;
7. correlation between CD8+ T-cells (as measured by standard flow cytometry) and the W1/W2 area on the XN WPC channel;

Exploratory:

Association of uncontrolled viral infection and the following as measured on the XN-20 platform

* % of lymphocytes mainly synthesizing antibodies with high fluorescence intensity (AS-Lymph);
* absolute and % lymphocytes reacting to infection with high fluorescence intensity (RE-Lymph);
* % reactive monocytes
* Neutrophil reactivity intensity;
* Neutrophil granularity intensity;
* Immature platelet fraction;
* Comparison of the blood film (DI-60 Review) and selected WBC subset read outs from the XN-20.
* Review of WDF lymphocyte cloud positional information using - HFLC/LY-X/LY-Y/LY-Z/LY-WX/LY-WY/LY-WZ.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years;
* Registered patient at Mortimer Market Centre;
* Willing to have a blood draw for the purpose of the study or, if the participant is having a blood draw for routine care, willing to have an additional EDTA sample taken at the time of that routine blood draw and willing that the results of the sample being drawn for standard care (FBC and T-cell subsets) can be used for this study;

In one of the four mutually exclusive groups:

i) Group A: HIV-infected (chronic or acute infection) with a HIV viral load of >1000 copies/mL in the 6 months prior to study entry and not (yet) in receipt of combination antiretroviral therapy (cART) at study entry; ii) Group B: HIV-infected on cART with HIV viral load <50 copies/mL within the 6 months prior to study entry, at least one measure of HCV (chronic or acute infection) showing a detectable HCV viral load and not in receipt of HCV treatment at study entry; iii) Group C: HCV mono-infected (chronic or acute infection) with detectable HCV viral load (>lower limit of quantification) in the prior 6 months and not in receipt of HCV treatment at study entry; iv) Group D: HBV mono-infected (chronic or acute infection) patients with detectable HBV viral load in the prior 6 months and not in receipt of HBV treatment at study entry.

- written informed consent.

Exclusion Criteria:

* On immunosuppressants and/or receiving chemotherapy or radiotherapy for a malignancy;
* Intercurrent infection within the prior 30 days (e.g. influenza like illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four groups of participants with chronic or acute viral infections :1) Group A: untreated Human Immunodeficiency Virus (HIV)-infected; 2) Group B: HIV-hepatitis C (HIV/HCV) coinfected, with treated HIV but untreated HCV; 3) Group C: untreated HCV monoinfection; 4) Group D: untreated Hepatitis B (HBV) monoinfection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-10-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of lymphocytes measured in area D1+D2 of the XN WDF and W1/W2 ratio from the WPC channel. | Day 1

SECONDARY OUTCOMES:
% lymphocytes in the D1 and D2 area of the XN WDF channel | Day 1
  as above
% lymphocytes in the D0 area of the XN WDF channel; | Day 1
  as above
correlation between CD4+ T-cells (as measured by standard flow cytometry) and the D1+D2 area on the XN WDF channel; | Day 1
  as above
correlation between CD8+ T-cells (as measured by standard flow cytometry) and the D1+D2 area on the XN WDF channel; | Day 1
  as above
correlation between CD4+ T-cells (as measured by standard flow cytometry) and the W1/W2 area on the XN WPC channel; | Day 1
  as above
correlation between CD8+ T-cells (as measured by standard flow cytometry) and the W1/W2 area on the XN WPC channel; | Day 1
  as above

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Pett, MD/PhD, Study Chair — University College, London
Locations (1):
- Mortimer Market centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We aim to recruit 100 participants in total, which will give us twenty-five participants per group. This is a convenience sample size that considered reasonable for this pilot, and can be recruited in the time frame allowed for this study, approximately 6 months. A simple descriptive analysis of data collected from the convenience sample will be presented. It is planned that results of this study will be published following its completion. There is no plan to inform participants of their individual data. The rationale for this is that this is an experimental testing platform, and it is unknown what the findings mean in the context of an individual participants' medical care. However, a letter summarising the group data will be developed and following approval by the IRB, given to all participants.